CLINICAL TRIAL: NCT00356161
Title: Open One-Arm Therapy Optimizing Trial on Regional Chemotherapy of the Liver Through an Interventionally Implanted A.Hepatica Port System in Patients With Liver Metastases or Primary Liver Neoplasms.
Brief Title: HAI Via Interventionally Implanted Port Catheter Systems
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVK-HAI 1
Record Dates: First submitted 2006-07-24; First posted 2006-07-25 (Estimated); Last update posted 2006-07-25 (Estimated); Status verified 2006-07

CONDITIONS: Colorectal Cancer; Liver Neoplasms; Hepatocellular Carcinoma; Gallbladder Cancer; Bile Duct Cancer
Keywords: colorectal neoplasms; hepatocellular carcinoma; gallbladder cancer; bile duct cancer; hepatic arterial infusion
MeSH Terms: conditions — Colorectal Neoplasms; Liver Neoplasms; Carcinoma, Hepatocellular; Gallbladder Neoplasms; Bile Duct Neoplasms

INTERVENTIONS:
Device: interventionally implanted hepatic arterial port catheter

SUMMARY:
Procedures to provide interventional implantation of a port catheter system into the hepatic artery and adjacent regional chemotherapy of the liver are optimized in the scope of an open, single-arm trial in patients with metastases and cancers confined to the liver. The primary objective is the improvement of indication, implantation procedure, and regional chemotherapy. Secondary objectives are port patency, comparison of complications with a historical collective of patients provided with a surgical hepatic arterial port device (colorectal cancer patients only), progression free and overall survival, efficacy of maintaining regional chemotherapy with 5-FU in combination with systemic treatment in patients with extrahepatic progression, quality of life.

DETAILED DESCRIPTION:
Inclusion criteria:

* histologically confirmed hepatic cancer without symptomatic extrahepatic manifestation.
* non-resectable disease or hepatic resection or ablation in between the past 8 weeks.
* measurable disease (at least before hepatic resection)
* Karnofsky performance status => 70%, or ECOG status 0-2
* >18 years of age
* life expectancy > 6 months
* compliance of the patient
* written informed consent

Exclusion criteria:

* second neoplasia within the past 3 years, except for non-melanotic skin cancer, adequately treated Ca in situ of cervix uteri, or adequately resected second colorectal cancer (in patients with liver metastases of colorectal cancer)
* symptomatic extrahepatic disease, in particular disseminated bone metastases, brain metastases
* liver cirrhosis with portal hypertension, active hepatitis B or C, previous percutaneous radiotherapy of the liver
* active infection
* history of gastric or duodenal ulcer
* symptomatic or uncontrolled peripheral arterial occlusive disease, history of stenosis of the renal artery.
* history of dilatative cardiomyopathy, vitium of mitral or aortic valve, persisting foramen ovale, atrial fibrillation
* artificial heart valve or vascular
* history of diabetic microangiopathy
* uncontrolled hyperthyriodism
* other severe concomitant disease (heart failure >NYHA 2°, respiratory failure, renal failure >stage2, liver failure (TPZ <50%).
* inherited or acquired immunodeficiency syndrome
* contraindication against 5-FU
* pregnancy and nursing, no contraception
* limited contractual capability.

After enrollment, an a port catheter catheter system is interventionally implanted into the hepatic artery and the patient is scheduled for regional chemotherapy according one out of 8 pre-defined chemotherapy schedules. All regimens are based on 5-fluorouracil and leucovorin, and optionally contain intraarterial mitomycin, oxaliplatin, or additional intravenous irinotecan.

Patients are followed up and evaluated for primary and secondary endpoints. After the inclusion of 50 patients treated and follow up at our institution, the study population has been extended to 100 patients in 8/2004.

ELIGIBILITY:
Inclusion Criteria:

see above

Exclusion Criteria:

see above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2002-04; Study Completion 2008-04

PRIMARY OUTCOMES:
Comparison of evaluation and intervention group
Complication rate (device implantation)
Safety of device and regional therapy

SECONDARY OUTCOMES:
prospective evaluation of port duration
comparison of complication and port duration with an historical collective of patients provided with a surgically implanted hepatic arterial port catheter system (liver metastases of colorectal cancer)
response
progression free and overall survival
efficacy of maintaining regional therapy combined with systemic chemotherapy in patients with extrahepatic progression while on study
quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Bert Hildebrandt, MD, Study Chair — Charté Centrum Tumormedizin, CVK, D-13344 Berlin; Hanno Riess, MD, PhD, Study Chair — Charité Centrum Tumormedizin, CVK, D-13344 Berlin; Jens Ricke, MD, PhD, Study Chair — Klinik für Radiologie und Nuklearmedizin, Universität Magdeburg, Leipziger Str. 44, D-39120 Magdeburg; Roland Felix, MD, PhD, Study Chair — Klinik für Strahlenheilkunde, CVK, Charité Universitätsmedizin Berlin, D-13344 Berlin; Peter Neuhaus, MD, PhD, Study Chair — Charité Centrum Chirurgische Medizin, CVK, D-13344 Berlin
Locations (2):
- Germany (2):
  - Charité Centrum Tumormedizin, Medizinische Klinik für Hämatologie und Onkologie, CVK, Berlin
  - Klinik für Radiologie und Nuklearmedizin, Otto-von-Guericke Universität Magdeburg, Magdeburg

REFERENCES:
- [Background] Ricke J, Hildebrandt B, Miersch A, Nicolaou A, Warschewske G, Teichgraber U, Lopez Hanninen E, Riess H, Felix R. Hepatic arterial port systems for treatment of liver metastases: factors affecting patency and adverse events. J Vasc Interv Radiol. 2004 Aug;15(8):825-33. doi: 10.1097/01.RVI.0000136992.96374.60. PMID 15297586